CLINICAL TRIAL: NCT02398565
Title: Pregnancy Subsequent to Ventral Hernia Repair: a Nationwide Cohort Study
Brief Title: Pregnancy Subsequent to Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Erling Oma, stud.med., Bispebjerg Hospital
Other Study IDs: BBH-2015-009
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Hernia, Ventral; Pregnancy
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients with a history of ventral hernia repair (umbilical/epigastric and incisional) with subsequent pregnancy
  Ventral hernia repair - perioperative factors of interest:
  - mesh vs sutured repair, age, planned vs emergency repair, open vs laparoscopic approach,
  Pregnancy and delivery - factors of interest:
  - vaginal vs caesearan section, single vs multiple pregnancy
  Subgroup of patients with mesh repair:
  - subanalysis on main attributes
  Subgroup of patients with sutured repair:
  - mono- vs multifilament, slowly vs rapidly absorbable
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
We will examine the outcome of ventral hernia repair with subsequent pregnancy

ELIGIBILITY:
Inclusion Criteria:

* History of ventral hernia repair with subsequent pregnancy
* Born between January 1 1955 and January 1 1995

Exclusion Criteria:

* Registered in the Danish Hernia Database with a non-valid ID-number, i.e. non-Danish resident.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nationwide study population of patients registered with a ventral hernia repair in The Danish Hernia Database between January 1 2007 and December 31 2014
Sampling Method: Non-Probability Sample
Enrollment: 7612 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Recurrence of ventral hernia | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars N Jorgensen, Study Chair — Bispebjerg Hospital
Locations (1):
- Digestive Disease Center, Bispebjerg Hospital, Copenhagen, Denmark